CLINICAL TRIAL: NCT04553341
Title: Induction of Cortical Plasticity by Navigated Transcranial Magnetic Stimulation
Brief Title: Induction of Cortical Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Sandro M. Krieg, apl. Prof. Dr. med. Sandro M. Krieg, MBA, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 404/18 S-AS
Record Dates: First submitted 2020-08-27; First posted 2020-09-17 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therepeutic (Experimental): rTMS
  Interventions: Device: Navigated repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Navigated repetitive transcranial magnetic stimulation — In these patients we will apply the following protocol: after the initial nTMS mapping of the according function, patients will be stimulated on 20 consecutive days by a series of rTMS pulses. The frequencies (1-20 Hz), number of pulses (100-1,000), and stimulation intensities (50-130% resting motor threshold = rMT = individual lowest stimulation intensity that evokes positive muscle responses) will be applied in dependency of the individual patients comfort and the evoked effect. Stimulations will be applied to the eloquent brain region, which is infiltrated by the tumor.

SUMMARY:
The study aims to induce plastic reorganization by a therapeutic protocol to increase the rate of gross total resection (GTR) and to optimize the oncological result.

DETAILED DESCRIPTION:
Regarding the therapy of cerebral parenchyma tumors, the extent of resection (EOR) has a significant impact on the prognosis. However, total resection is not possible in up to 65% of cases because these tumors frequently infiltrate eloquent areas such as language or motor centers. Consequently, an optimal oncologic result from the surgical perspective cannot be achieved in a considerable large amount of patients. One possible solution is based on the tumor-induced shift of functional areas, which can move away from their original localization. Earlier studies already described the resection of glioma residuals during a second surgery after plastic reorganization has taken place. The authors complained that this reorganization is not detectable without surgery. Navigated transcranial magnetic stimulation (nTMS) was developed for the noninvasive localization of motor and language areas, which enables us to detect the spatial shift of cortical motor and language functions in tumor patients. Recent publications were already able to demonstrate that the individual and exact localization of the motor cortex leads to an increased EOR and prolongs the progression-free survival (PFS). Therefore, the current project intends to take advantage of this plastic reorganization for EOR optimization in cerebral parenchyma tumors. In this context, nTMS is supposed to also induce this plasticity within the frame of a repetitive stimulation protocol (rTMS). Besides other therapeutic applications, rTMS also showed a positive effect on the improvement of aphasia as well as motor recovery in patients after stroke, even in randomized multicenter studies, by inducing plastic reorganization. Moreover, rather than waiting for tumor-induced plastic reorganization, the investigators also aim to use the potential of rTMS for spatial plastic reorganization of functional areas adjacent to intracerebral parenchymal tumors to move functionally eloquent brain regions away from the planned resection cavity.

ELIGIBILITY:
Inclusion Criteria:

* Intracerebral tumor
* Cortical function is located within planned resection area as confirmed by preoperative navigated transcranial magnetic stimulation and/or intraoperative direct electrical stimulation mapping
* Informed consent for participation
* Age >18 years

Exclusion Criteria:

* Prognosis less than 6 months
* Contraindications for MRI or nTMS (cardiac pacemaker, deep brain stimulator, cochlea implant
* Karnofsky-performance-index <60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Cortical location of function (nTMS) | 3 months
  Location of cortical motor or language function as measured by navigated transcranial magnetic stimulation (nTMS) mapping

SECONDARY OUTCOMES:
Cortical location of function (rsfMRI) | 3 months
  Location of cortical motor or language function as measured by resting state functional MRI (rsfMRI)
Cortical location of function (DES) | 3 months
  Location of cortical motor or language function as measured by intraoperative direct electrical stimulation (DES)
Cortical location of function (nTMS / rsfMRI / DES) | 6 months
  Location of cortical motor or language function as measured by nTMS, rsfMRI, and /or DES
Cortical location of function (nTMS / rsfMRI / DES) | 9 months
  Location of cortical motor or language function as measured by nTMS, rsfMRI, and /or DES
Cortical location of function (nTMS / rsfMRI / DES) | 12 months
  Location of cortical motor or language function as measured by nTMS, rsfMRI, and /or DES

CONTACTS AND LOCATIONS:
Overall Officials: Sandro M Krieg, MD, MBA, Principal Investigator — Technical University of Munich
Locations (1):
- Department of Neurosurgery, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
After confirmation by the local ethics committee, individual participant data that underlie the results reported in the manuscript will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol
Time Frame: Data will be available after deidentification, beginning nine months and ending 36 months following article publication.
Access Criteria: Data will be available for individual participant data meta-analysis. Requestors will need to sign a data access agreement. Information regarding submitting proposals and accessing data will be published. Data will be made available by contacting the corresponding author of this manuscript via email.